CLINICAL TRIAL: NCT06984523
Title: A Phase II Single-Arm Study of Craniospinal Irradiation With Linac Based Volumetric Modulated Arc Therapy (VMAT) for Patients With Leptomeningeal Metastasis
Brief Title: Study of Craniospinal Irradiation With Linac Based Volumetric Modulated Arc Therapy (VMAT) for Patients With Leptomeningeal Metastasis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-01730
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Leptomeningeal Metastasis
MeSH Terms: conditions — Meningeal Carcinomatosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Linac based Volumetric Arc Therapy (VMAT) CSI (Experimental): Radiation dose will be administered according to the physician's written directive. Treatment will be administered once a day, Monday through Friday, for a total of ten fractions.
  Interventions: Radiation: Varian Eclipse

INTERVENTIONS:
Radiation: Varian Eclipse — Varian TrueBeam linear accelerator with photon beam Volumetric Modulated Arc Therapy (VMAT) capability. Subjects will receive 3000 centigray (cGy) in 10 fractions at 300 cGy per fraction.

SUMMARY:
The purpose of this study is to confirm the safety and efficacy of linac based Volumetric Modulated Arc Therapy (VMAT) for craniospinal irradiation (CSI) in solid tumor cancer patients with leptomeningeal metastasis. The primary aim is to determine if linac based VMAT CSI for leptomeningeal metastasis improves central nervous system (CNS) progression free survival (PFS) compared to the historical standard control CNS PFS in patients treated with Involved Field Radiation Therapy (IFRT).

ELIGIBILITY:
Inclusion Criteria:

1. Solid tumor cancer primary with leptomeningeal metastases established radiographically and/or by CSF cytology
2. Candidate for radiation therapy for the treatment of leptomeningeal metastases
3. If patient had prior radiation, a treatment plan can be generated that will not exceed normal tissue tolerances
4. Patient must have reasonable systemic treatment options, as confirmed by their medical oncologist
5. Age ≥ 18 years old
6. Able to provide informed consent
7. Karnofsky Performance Scale (KPS) ≥ 60
8. Adequate hematologic baseline

   1. Hemoglobin > 8g/dL
   2. Absolute neutrophil count >1,000/mm3
   3. Platelet count > 100,000/mm3
9. Female subjects must either be of

   1. Non-reproductive potential (over 60 years old, or without menses for at least 1 year without an alternative medical cause)
   2. Have history of hysterectomy, bilateral tubal ligation, or bilateral oophorectomy
   3. Must have negative serum/urine pregnancy test
   4. If of reproductive age, must practice effective contraceptive method

Exclusion Criteria:

1. Patient has multiple severe neurologic deficits per physician assessment
2. Patient has diffuse systemic disease without reasonable systemic therapy options
3. Patient is unable to undergo MRI brain and spine with gadolinium contrast
4. Prior radiation that would preclude development of a treatment plan that respects normal tissue constraints
5. Pregnant or lactating women
6. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-14 (Estimated); Primary Completion 2028-05-12 (Estimated); Study Completion 2028-05-12 (Estimated)

PRIMARY OUTCOMES:
Time to central nervous system (CNS) progression free survival | From baseline up to 1 year from end of treatment
  Time to CNS progression free survival will be estimated using Kaplan Meier methods for censored data that includes CNS progressions. CNS disease progression will be defined as new or worsening neurologic deficit unrelated to therapeutic intervention via neurological assessment using Neurologic Assessment in Neuro-Oncology (NANO) scale, cerebrospinal fluid (CSF) cytology being newly positive for malignancy after initially being negative, MRI brain with and without contrast or MRI total spine with and without contrast shows progression per the European Organization for Research and Treatment of Cancer (EORTC) Brain Tumor Group and the Response Assessment in Neuro-Oncology (RANO) scorecard.

SECONDARY OUTCOMES:
Overall survival | From baseline up to 1 year from end of treatment
  Overall survival will be estimated using Kaplan Meier methods for censored data that includes deaths as events.
Time to CNS progression | From baseline up to 1 year from end of treatment
  Time to CNS progression will be analyzed using competing risk methods, considering death and progression from other causes as competing risks.
Rate of cessation of systemic therapy | 1 year post-treatment
Number of treatment-related adverse events | End of study (up to 2 years)
M.D. Anderson Symptom Inventory - Brain Tumor (MDASI-BT) score | End of study (up to 2 years)
  The MDASI-BT includes 22 items assessing severity of brain tumor symptoms and 6 items assessing interference. Symptom severity and interference are assessed on a scale from 0-10 scale. A score of 0 indicates "not present" or "did not interfere," while a score of 10 represents "as bad as you can imagine" or "interfered completely". Scores range from 0-280. Higher scores indicate the brain tumor significantly impairs daily functioning.
M. D. Anderson Symptom Inventory - Spine Tumor (MDASI-SP) score | End of study (up to 2 years)
  The MDASI-SP includes 18 items assessing severity spinal tumor symptoms and 6 items assessing interference. Symptom severity and interference are assessed on a scale from 0-10 scale. A score of 0 indicates "not present" or "did not interfere," while a score of 10 represents "as bad as you can imagine" or "interfered completely". Scores range from 0-240. Higher scores indicate the brain tumor significantly impairs daily functioning.
Functional Assessment of Cancer Therapy - Brain (FACT-Br) score | End of study (up to 2 years)
  The FACT-Brain (FACT-Br) is one such instrument that assesses brain-tumor related QOL issues. The questionnaire consists of the FACT-G plus a brain-tumor specific scale. A total of 50 items are included that cover the following domains of QOL: physical well-being, social/family well-being, emotional well-being, functional well-being, and disease specific concerns. Patients are asked to indicate the presence/severity of certain issues/symptoms on a scale of 0 - 4 (a 5-point Likert Scale). Higher scores indicate decreased health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Cooper, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Benjamin.cooper@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Benjamin.cooper@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.